CLINICAL TRIAL: NCT06634511
Title: Core Stability Exercise Versus Aerobic Exercise on Pain, Range of Motion and Function in Patients With Chronic Mechanical Low Back Pain: Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeinab Abd el fattah Ali, assistant professor of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-96
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Patients With Chronic Mechanical LBP
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core stability exercise group (Experimental): Group A: core stability exercise group:15 Patients assigned to this group will undergo a core stability exercises.2times per week /8weeks.in addition to traditional physical therapy program
  Interventions: Other: core stability exercises
- aerobic exercise group (Experimental): Group B:(aerobic exercise group) 15 patients will receive aerobic exercise in the form of treadmill for 30 minutes2 session per week/8 weeks
  Interventions: Other: core stability exercises
- traditional physical therapy group (Experimental): Group C(conventional group): 15 patients will receive Infrared radiation (using BL 220 Infrared lamp, MT03009201 model) for 15 minutes, Transcutaneous Electrical Nerve stimulation (using model DX66053, pain modulation mode) for 10 minutes, Participants were treated twice weekly
  Interventions: Other: core stability exercises

INTERVENTIONS:
Other: core stability exercises — Group A: core stability exercise group:15 Patients assigned to this group will undergo a core stability exercises" ts.2times per week /8weeksin addition to conventional therapy (Infrared radiation (using BL 220 Infrared lamp, MT03009201 model) for 15 minutes, Transcutaneous Electrical Nerve stimulation (using model DX66053, pain modulation mode) for 10 minutes
  Group B:(aerobic exercise group) 15 patients will receive aerobic exercise in the form of treadmill for 30 minutes2 session per week/8 weeks
  Group C(conventional group): 15 patients will receive Infrared radiation (using BL 220 Infrared lamp, MT03009201 model) for 15 minutes, Transcutaneous Electrical Nerve stimulation (using model DX66053, pain modulation mode) for 10 minutes, Participants were treated twice weekly
  Other Names: aerobic exercise

SUMMARY:
Chronic mechanical low back pain (CMLBP) is a prevalent musculoskeletal condition characterized by persistent pain originating from the spine, muscles, ligaments, or intervertebral discs. It is one of the leading causes of disability worldwide. (CMLBP) have significantly affected the individual's physical, emotional, and social well-being, as well as their overall quality of life, functional capacity, and productivity of individuals. Unlike acute low back pain, which typically resolves within a few weeks, CMLBP persists for more than three months and often fluctuates in intensity, leading to recurrent episodes of pain and discomfort [1]. Chronic mechanical low back pain (LBP) has been the subject of extensive research, with numerous studies highlighting its multifactorial nature and varied treatment outcomes. Previous research has established that chronic mechanical LBP often results from prolonged strain on the lumbar spine due to poor posture, repetitive stress, or underlying musculoskeletal imbalances. Studies have consistently shown that interventions such as physical therapy, which includes strengthening exercises and ergonomic adjustments, can be effective in alleviating symptoms and improving functional outcomes.

However, evidence also suggests that the efficacy of these treatments can be limited by factors such as patient adherence and the presence of psychological components like anxiety and depression.

Furthermore, recent research emphasizes the importance of a multidisciplinary approach that integrates both physical and psychological therapies to address the complex nature of chronic mechanical LBP more comprehensively [2]. Aerobic exercise involves activities that increase the heart rate and improve cardiovascular endurance. The rationale for using aerobic exercise in the management of CMLBP is based on several physiological mechanisms. Firstly, aerobic exercise enhances blood ow and nutrient delivery to the spine and surrounding musculature, which can promote healing and reduce muscle stiffness.

Secondly, regular aerobic activity has been shown to reduce systemic inflammation and increase endorphin production, both of which can lower pain perception. Additionally, aerobic exercise can improve psychological well-being, which is an important factor given the strong association between chronic pain and mental health conditions like depression and anxiety [1]. Core stability training focuses on strengthening the muscles that support the spine, including the transversus abdominis, multifidus, pelvic floor muscles, and other muscles of the abdomen, lower back, and pelvis. These muscles play a critical role in maintaining spinal stability and proper alignment, which is essential for preventing and managing back pain. Core stability exercises, such as planks, bridges, and lumbar stabilization exercises, aim to enhance the endurance and coordination of these muscles, thereby reducing excessive spinal movements and mechanical strain that can exacerbate pain [3] Aerobic exercise and core stability training are commonly recommended for chronic mechanical low back pain (CMLBP). but to our knowledge, there is insufficient evidence comparing the relative effectiveness of aerobic exercise and core stability training, leaving a gap in understanding which approach provides superior outcomes for CMLBP. So the aim of our study is to compare between the effectiveness of aerobic exercise and core stability training on pain, range of motion, flexibility, and functional abilities in patients of CMLBP.

DETAILED DESCRIPTION:
Study Design:

Randomized control trail study. 2.2. Study Area: Faculty of applied medical sciences, physiotherapy department at Jouf University 2.3. Study Population: We will include studies that evaluated patients over 18years of age and below 50 years with chronic non-specific low back pain defined as pain or discomfort lasting more than 12weeks in the region below the last costal margins and above the lower gluteal folds, without symptoms in the lower limbs [4].. 2.3.1. Inclusion Criteria: All females between 18-50 years have mechanical LBP more than 3 months 2.3.2. Exclusion Criteria: Patients will be excluded if they evaluated patients with nerve root compromise, metabolic or serious spinal pathologies (e.g., fractures, tumors, inflammatory, and infectious diseases), previous spinal surgery, postpartum low back pain or pelvic pain due to pregnancy, and pain unrelated to the lower back.

Assessment tools:

Numerical rating scale:

Pain Numeric Rating Scale (PNRS): The PNRS is a straightforward tool where patients rate their pain on a scale from 0 (no pain) to 10 (worst possible pain).

It provides a subjective measure of pain intensity and is widely used due to its simplicity and effectiveness in capturing a patient's perceived pain level, Pain scores were classified as follows: 0 (no pain), 1-3 (mild), 4-7 (moderate), and 8-10 (high) [5].

Range of Motion (ROM):

Lumber ROM will be assessed by A standard gravity-based inclinometer (model A-300; Vertex Co., Taiwan) for assessing flexion, extension and lateral bending

Modified modified schober test for assessment of lumber flexibility: Modified Modified Schober Test (MMST)is a modification of Modified Schober Test(MST) by Van Adrichen and Van der Korst(1973). It uses two marks one over the spine connecting two PSIS and other over 15 cm superior to first mark. It eliminates the errors in identification of lumbosacral junction and make sure that entire lumbarspine was included. [6]

The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluatorsFAIRS & RESEARCH CENTER use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools [7].

ELIGIBILITY:
Inclusion Criteria:

* All females between 18-45 years have mechanical LBP more than 3 months

Exclusion Criteria:

* Patients will be excluded if they evaluated patients with nerve root compromise, metabolic or serious spinal pathologies (e.g., fractures, tumors, inflammatory, and infectious diseases), previous spinal surgery, postpartum low back pain or pelvic pain due to pregnancy, and pain unrelated to the lower back.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale: | 1 month
  ain Numeric Rating Scale (PNRS): The PNRS is a straightforward tool where patients rate their pain on a scale from 0 (no pain) to 10 (worst possible pain).
  It provides a subjective measure of pain intensity and is widely used due to its simplicity and effectiveness in capturing a patient's perceived pain level,
Range of motion Range of Motion (ROM): Range of Motion (ROM): | 1 month
  Lumber ROM will be assessed by A standard gravity-based inclinometer (model A-300; Vertex Co., Taiwan) for assessing flexion, extension and lateral bending
Modified modified schober test for assessment of lumber flexibility: | 1 month
  Modified Modified Schober Test (MMST)is a modification of Modified Schober Test(MST) by Van Adrichen and Van der Korst(1973). It uses two marks one over the spine connecting two PSIS and other over 15 cm superior to first mark. It eliminates the errors in identification of lumbosacral junction and make sure that entire lumbarspine was included.

SECONDARY OUTCOMES:
The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) | 1 month
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools .

CONTACTS AND LOCATIONS:
Locations (1):
- Jouf university, Qurayyat, Jouf, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No